CLINICAL TRIAL: NCT02799576
Title: A Curved Block Needle for the Infraclavicular Brachial Plexus Block in Patients Undergoing Surgery Distal to the Elbow
Brief Title: A Curved Block Needle for the Infraclavicular Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Tarek F.Tammam, Prof. of anesthesia and intensive care,faculty of medicine,Suez Canal University, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TFTammam; Ghada A. K (Other: Suez Canal University)
Record Dates: First submitted 2016-06-06; First posted 2016-06-15 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Needle Track
Keywords: Ultrasound; Regional blockade; Infraclavicular brachial plexus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curved needle (Experimental): This will utilize the curved block needle of performance of regional block
  Interventions: Device: Curved needle
- Traditional needle (No Intervention): This will utilize the traditional block needle of performance of regional block

INTERVENTIONS:
Device: Curved needle — In this arm, the curved block needle will be used for regional blockade
  Arms: Curved needle

SUMMARY:
The investigators hypothesized that using the curved needle could facilitate the block placement and provide short procedure time. Aim of the work: The investigators will compare namely straight and curved block needle with in-plane needle insertion techniques for the infraclavicular brachial plexus nerve block (ICNB) regarding the block performance time.

DETAILED DESCRIPTION:
Sometimes, there is a limited block needle access at the inferior edge of the clavicle while performing in- plane infraclavicular parasagittal blockade. This might present a challenge in manipulating and visualizing the block needle in easy way along its entire trajectory during the blockade. The curved block needle might have its positive impact on the capacity to control the block needle advancement relative to the target nerve.

70 patients between the ages of 18 and 60 years with American Society of Anesthesiologists (ASA) physical status I- II, scheduled for elective surgery distal to the elbow will be enrolled in a prospective, comparative, randomized clinical study.

Patients will be randomly assigned into two groups: C (n = 35), in whom US-guided single injection ICNB will be performed using a curved line needle; and S (n = 35), in whom US-guided ICNB will be performed using a straight line needle. All patients will be pre-medicated with oral diazepam (7.5 mg) 30 min before the procedure, and IV fentanyl (50 ug) will be administered 5 minutes before placement of the block. Before the procedure, an IV access and standard monitoring of electrocardiogram (ECG), noninvasive blood pressure (NIBP), and peripheral oxygen saturation (SPO2) will be established.

The ultrasound guided Infraclavicular brachial plexus block will be performed in the block room using a linear-array US probe (8-13 MHz). The ultrasound probe will be placed just below the lower edge of the clavicle and medial to the coracoid process (parasagittal orientation), with adjustment of depth, frequency and gain to spot the best view of the transverse axillary artery and its surrounding cords (short-axis view).

After sterile skin preparation with chlorhexidine solution, local infiltration with 2 ml of lidocaine (10 mg/ml) will be made at the cephalad aspect of the ultrasound probe. A 10-cm, short-bevel block (straight or curved) needle will be attached to the nerve stimulator delivering a current of 1.2 mA ( milliampere) at a frequency of 2 Hz (Hertz), will be inserted in-plane just inferior to the clavicle.

After eliciting the posterior cord motor response (finger or wrist extension) with a current intensity of ≤ 0.5 mA, correct needle-tip position will be confirmed by test injections with 1 ml of 5 % dextrose solution. Then, thirty milliliters of local anesthetic mixture (lidocaine 10 mg/ml and bupivacaine 2.5 mg/ml) will be incrementally injected after careful aspiration. The goal is to ensuring a U-shaped distribution of anaesthetic solution with anterior displacement of the axillary artery.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 60 year old both sex, able to provide informed consent to participate, enrolled in elective surgery distal to the elbow, single procedure.

Exclusion Criteria:

* Unable to consent to participate, known to have lidocaine or bupivacaine allergy, more than one procedure will be performed at the same setting, patients with local infections,neuropathies, coagulopathies,and history of chronic analgesic therapy, Obesity (body mass index ≥ 30 kg/m2),

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Performance time | 12 min
  The time to perform the Infraclavicular brachial nerve block. Performance time is defined as the sum of recognition time and local anesthetics injection time. Recognition time is defined as the time interval in seconds (s) from needle insertion to achievement of proper motor response. Local anesthetics injection time is defined as the time interval in seconds (s) between the achievement of motor response and the end of local anesthetics injection through the block needle

SECONDARY OUTCOMES:
Number of needle attempts to elicit proper motor response | 12 min
  New attempt will be defined as needle reinsertions through separate skin puncture.
Number of needle redirections to elicit proper motor response | 12 min
  Needle redirection will be defined as draw back and redirects the needle if no proper nerve response could be elicited.
The Infraclavicular brachial nerve block success rate | 30 min after local anesthetics administration
  The Infraclavicular brachial nerve block success will be assessed according to the adequacy of surgical anesthesia and is defined as complete loss of pinprick sensation within 30 min of anesthetic administration and if no supplementation (sedative or analgesic) is required during surgery. Partial block is defined as inadequate sensory blockade after 30 min of anesthetic administration. The supplementation (IV analgesic, rescue blocks or local infiltration) is required to complete the proposed surgery. Failed block is considered if general anesthesia is required to complete the proposed surgery.
Patient satisfaction | during surgical procedures
  All patients will be asked to rate their discomfort during the block placement and tourniquet pain using the Verbal Rating Scale (VRS: 0 = no discomfort, 10 = the worst discomfort).
Anesthesiologist satisfaction | 12 min
  Level of anesthesiologist satisfaction for using different block needles will be evaluated using VRS (0, no satisfaction; 10, maximum satisfaction).

OTHER OUTCOMES:
Incidence of adverse events | Intraoperative and in the first 48 post-operative hours
  Incidence of adverse events and complications during and after the procedure will be also recorded. Complications, including hematoma, infection and neuropathies, will be recorded intraoperatively and in the first 48 post-operative hours.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek F. Tammam, Prof., Study Director — Suez Canal university,Faculty of Medicine
Locations (1):
- Suez canal University hospital, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tammam TF, Kamhawy GA. Use of a curved needle to facilitate lateral sagittal infraclavicular block performance: a randomized clinical trial. J Anesth. 2019 Oct;33(5):604-611. doi: 10.1007/s00540-019-02674-w. Epub 2019 Aug 29. PMID 31468177